CLINICAL TRIAL: NCT05542173
Title: National, Multicenter, Randomized, Double-blind, Phase III Clinical Trial to Evaluate the Efficacy and Safety of BALI Association in the Treatment of Aphthous Ulcerations
Brief Title: Efficacy and Safety of BALI Association in the Treatment of Aphthous Ulcerations
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0322 - BALI
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Aphthous Stomatitis
Keywords: Aphthous Stomatitis
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BALI 25 + 25 + 15 (Experimental): Three applications per day or more in case of pain, not exceeding six applications per day. The number of drops varies according to the ulcer diameter: 1 to 3 mm: 1 drop; 3 to 6 mm: 2 drops; greater than 6 mm: 3 drops.
  Interventions: Drug: BALI association
- PLACEBO (Placebo Comparator): Three applications per day or more in case of pain, not exceeding six applications per day. The number of drops varies according to the ulcer diameter: 1 to 3 mm: 1 drop; 3 to 6 mm: 2 drops; greater than 6 mm: 3 drops.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BALI association — BALI association oral suspension, 25 mg + 25 mg + 15 mg, oral. Three applications per day or more in case of pain, not exceeding six applications per day.
  Arms: BALI 25 + 25 + 15
Drug: Placebo — Placebo. Three applications per day or more in case of pain, not exceeding six applications per day.
  Arms: PLACEBO

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of BALI association in the treatment of aphthous ulceration.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Age greater than or equal to 12 years;
* Minor recurrent aphthous ulceration with onset of symptoms within 48 hours;
* Moderate to severe baseline pain, with VAS ≥ 4 (EVA scale).

Exclusion Criteria:

* Any clinical findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* Participants diagnosed with: Behcet's disease, rheumatoid arthritis, systemic lupus erythematosus, reactive arthritis, Reiter's syndrome, Crohn's disease, ulcerative colitis);
* Participants with diseases that affect healing (e.g. diabetes);
* Immunocompromised participants;
* Participants with aphthous herpetiform ulceration or major aphthous ulceration;
* Participants using medication to treat oral ulcerations (systemic or local);
* Participants who used analgesics or anti-inflammatory drugs in the 6 hours prior to the beginning of the study;
* Participants who used systemic antibiotics in the 2 weeks prior to the beginning of the study;
* Participants using medications that can confuse pain assessment (psychotropics, antidepressants and sedative-hypnotics), except when on a stable dose for at least 30 days prior to the screening visit, and the dose cannot be changed during the clinical trial;
* Participants with current smoking habits.
* Participants who are pregnant, breastfeeding or planning to get pregnant or female participants with the potential to become pregnant who are not using a reliable method of contraception;
* Known hypersensitivity to the formula components used during the clinical trial;
* Participants with current or medical history of cancer in the last 5 years;
* Participants who participated in other research protocol in the last 12 months, unless the investigator judges that there may be a direct benefit to it.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
To assess the reduction in pain intensity after 3 days of treatment. | 3 days
  Difference in pain intensity after 3 days of treatment compared to baseline. Pain intensity will be evaluated by the Visual Analogue Scale (VAS). The VAS consists of a 10 cm line, with two end points representing 0 ("no pain") and 10 (pain as bad as it could possibly be").

SECONDARY OUTCOMES:
To assess the reduction in pain intensity after the first application. | 15 minutes
  Difference in pain intensity 15 minutes after the first application of the medication compared to baseline, measured by the VAS scale. The VAS consists of a 10 cm line, with two end points representing 0 ("no pain") and 10 (pain as bad as it could possibly be").
To assess the reduction in pain intensity during the treatment. | 5 and 7 days
  Difference in pain intensity after 5 and 7 days of treatment compared to baseline, measured by the VAS scale. The VAS consists of a 10 cm line, with two end points representing 0 ("no pain") and 10 (pain as bad as it could possibly be").
Percentage of participants healed during treatment. | 3, 5 and 7 days
  Percentage of participants healed after 3, 5, and 7 days of treatment, defined as ulcer diameter = 0 mm and pain intensity = 0, measured by the Likert scale. Likert scale is a five point scale: 0 = no pain and 4 = pain as bad as it could possibly be".
Percentage of participants with no pain during treatment. | 3, 5 and 7 days
  Percentage of participants with no pain after 3, 5, and 7 days of treatment, measured by the Likert scale. Likert scale is a five point scale: 0 = "no pain" and 4 = "pain as bad as it could possibly be".
To assess the percentage change in pain intensity from baseline during treatment. | 3, 5 and 7 days
  Pain intensity will be evaluated by the VAS scale.The following calculations will be performed: ((D3, D5 or D7 - V0) / baseline) ×100%. The VAS consists of a 10 cm line, with two end points representing 0 ("no pain") and 10 (pain as bad as it could possibly be").

CONTACTS AND LOCATIONS:
Locations (1):
- EMS, Hortolândia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No